CLINICAL TRIAL: NCT01030718
Title: A Study to Document the Long-Term Safety and Efficacy of BMS-354825 in Subjects With Imatinib Resistant or Intolerant Chronic Myelogenous Leukemia and Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia Who Are Resistant or Intolerant to Previous Treatment and Have Completed the Previous Phase I/II Protocol (CA180-031/NCT00337454)
Brief Title: Rollover Study of BMS-354825 in Patients With CML and Ph+ALL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA180-036
Record Dates: First submitted 2009-12-10; First posted 2009-12-11 (Estimated); Results first posted 2010-12-14 (Estimated); Last update posted 2010-12-14 (Estimated); Status verified 2010-11

CONDITIONS: Chronic Myelogenous Leukemia; Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- dasatinib (CML-CP) (Experimental): CML - Chronic Phase
  Interventions: Drug: dasatinib
- dasatinib (CML-AP/BP) (Experimental): CML - Accelerated Phase and Blast Phase
  Interventions: Drug: dasatinib
- dasatinib (Ph+ ALL) (Experimental): Ph+ Acute Lymphoblastic Leukemia
  Interventions: Drug: dasatinib

INTERVENTIONS:
Drug: dasatinib — Tablet, Oral, (50mg, 70mg or 90mg BID on a continuous daily dosing schedule), allowed to modify within the range of 50 mg twice daily (BID) to 90 mg BID
  Other Names: Sprycel; BMS-354825

SUMMARY:
To assess the safety of dasatinib (BMS-354825) in subjects with Imatinib resistant or intolerant chronic myelogenous leukemia (CML) and Philadelphia chromosome positive (Ph+) acute lymphoblastic leukemia (ALL) who are resistant or intolerant to treatment and will continue study drug after completing the previous Phase I/II study (CA180031/NCT00337454)

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were eligible and completed the previous Phase I and II study (CA180031/NCT00337454) and for whom the principal investigator has deemed that continuation of study drug is in the best interest of the subject

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Subjects who are eligible and willing to undergo transplantation at pre-study
* Non-hematologic intolerance to Dasatinib (BMS-354825) in the previous Phase I and II study (CA180031/NCT00337454)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: CA180-031 = NCT00337454; CA180-036 = NCT01030718
Pre-assignment Details: 55 participants were randomized to study CA180-031; 1 participant with chronic myelogenous leukemia-chronic phase (CML-CP) was withdrawn prior to dosing due to thrombocytopenia. 54 subjects were treated; 44 subjects finished the study period of CA180-031 and transferred CA180-036. Analyses were done on the population enrolled into CA180-031 study.
Groups:
- CML - Chronic Phase (CML-CP): Imatinib resistant or intolerant CML-CP disease cohort who had completed the previous study (CA180031) phase I/II. The study drug was administered twice daily (BID). The starting dose level for this trial in each individual participant was the same dose level at the end of CA180031(ie, 50mg, 70mg or 90mg BID on a continuous daily dosing schedule), allowed to modify within the range of 50 mg twice daily (BID) to 90 mg BID.
- CML - Accelerated Phase and Blast Phase (CML-AP/BP): Imatinib resistant or intolerant CML-AP/BP disease cohort who had completed the previous study (CA180031) phase II. The study drug was administered twice daily (BID). The starting dose level for this trial in each individual participant was the same dose level at the end of CA180031 (ie, 50mg, 70mg or 90mg BID on a continuous daily dosing schedule), allowed to modify within the range of 50 mg twice daily (BID) to 90 mg BID.
- Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL): Philadelphia chromosome positive (Ph+) ALL subjects with resistance or intolerance to past therapy and who had completed the previous study (CA180031) phase II. The study drug was administered twice daily (BID). The starting dose level for this trial in each individual participant was the same dose level at the end of CA180031 (ie, 50mg, 70mg or 90mg BID on a continuous daily dosing schedule), allowed to modify within the range of 50 mg twice daily (BID) to 90 mg BID.
Period: Studies CA180-031 and -036 Combined
Arm/Group | CML - Chronic Phase (CML-CP) | CML - Accelerated Phase and Blast Phase (CML-AP/BP) | Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL)
Started | 30 | 11 | 13
Completed | 26 | 2 | 1
Not Completed | 4 | 9 | 12
Not completed — Insufficient effect | 1 | 1 | 11
Not completed — Adverse Event | 3 | 5 | 1
Not completed — Death | 0 | 1 | 0
Not completed — other reasons | 0 | 2 | 0
Period: Study CA180-036 Only
Arm/Group | CML - Chronic Phase (CML-CP) | CML - Accelerated Phase and Blast Phase (CML-AP/BP) | Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL)
Started | 29 | 9 | 6
Completed | 26 | 2 | 1
Not Completed | 3 | 7 | 5
Not completed — insufficient effect | 1 | 1 | 5
Not completed — Adverse Event | 2 | 3 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Other Reasons | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- CML - Chronic Phase (CML-CP): Imatinib resistant or intolerant CML-CP disease cohort who had completed the previous study (CA180031/NCT00337454) phase I/II. The study drug was administered twice daily (BID). The starting dose level for this trial in each individual participant was the same dose level at the end of CA180031(ie, 50mg, 70mg or 90mg BID on a continuous daily dosing schedule), allowed to modify within the range of 50 mg twice daily (BID) to 90 mg BID.
- CML - Accelerated Phase and Blast Phase (CML-AP/BP): Imatinib resistant or intolerant CML-AP/BP disease cohort who had completed the previous study (CA180031/NCT00337454) phase II. The study drug was administered twice daily (BID). The starting dose level for this trial in each individual participant was the same dose level at the end of CA180031 (ie, 50mg, 70mg or 90mg BID on a continuous daily dosing schedule), allowed to modify within the range of 50 mg twice daily (BID) to 90 mg BID.
- Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL): Ph+ ALL subjects with resistance or intolerance to past therapy and who had completed the previous study (CA180031/NCT00337454) phase II. The study drug was administered twice daily (BID). The starting dose level for this trial in each individual participant was the same dose level at the end of CA180031 (ie, 50mg, 70mg or 90mg BID on a continuous daily dosing schedule), allowed to modify within the range of 50 mg twice daily (BID) to 90 mg BID.
- Total: Total of all reporting groups
Arm/Group | CML - Chronic Phase (CML-CP) | CML - Accelerated Phase and Blast Phase (CML-AP/BP) | Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL) | Total
Number analyzed (Participants) | 30 | 11 | 13 | 54
Age, Customized [Number; unit: participants]
  <65 years | 26 | 8 | 10 | 44
  >=65 years | 4 | 3 | 3 | 10
Age Continuous [Median (Full Range); unit: years] | 51.5 [27 to 68] | 57.0 [31 to 73] | 64.0 [29 to 70] | 55.5 [27 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 6 | 19
  Male | 21 | 7 | 7 | 35
Region of Enrollment [Number; unit: participants]
  Japan | 30 | 11 | 13 | 54
Eastern Oncology Cooperative Group Performance Status [Number; unit: participants] — ECOG PS scale is a 6-item scale to assess disease progression, daily functioning, and appropriate treatment and prognosis. Scale=0-5, with 0=fully active, 1=restricted in physically strenuous activity but ambulatory, 2=ambulatory and capable of all selfcare but unable to work, 3= limited selfcare ability and confined to bed/chair >50% of waking hours, 4=completely disabled and no selfcare ability and confined to bed/chair, and 5=death
  participants
    Status = 0 | 27 | 6 | 9 | 42
    Status = 1 | 3 | 5 | 4 | 12
    Status = 2 | 0 | 0 | 0 | 0
    Status = 3 | 0 | 0 | 0 | 0
    Status = 4 | 0 | 0 | 0 | 0
    Status = 5 | 0 | 0 | 0 | 0
Imatinib Status [Number; unit: participants] — Resistance to Imatinib=Previously been treated with imatinib at a dose of ≥ 400 mg/day AND developed progressive disease while receiving imatinib at that dose. Intolerance to Imatinib=A subject is defined as being intolerant to imatinib if he or she had a Grade ≥3 toxicity considered at least possibly related to imatinib at a dose of ≤400 mg/day which led to discontinuation of therapy.
  participants
    Resistant | 18 | 8 | 9 | 35
    Intolerant | 12 | 3 | 4 | 19
Body Weight [Median (Full Range); unit: kg] | 64.05 [44.0 to 86.5] | 58.00 [43.6 to 76.6] | 53.20 [37.0 to 77.8] | 60.55 [37.0 to 86.5]
Height [Median (Full Range); unit: cm] | 163.65 [147.0 to 180.3] | 161.00 [145.7 to 174.5] | 164.50 [151.7 to 171.7] | 163.25 [145.7 to 180.3]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Deaths, and Discontinuation
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with this treatment. Related AE=relationship of certain, probable, possible, or missing. SAE=any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in development of drug dependency or drug abuse, is an important medical event.
Time Frame: baseline; every 4 weeks (if on study < 6 months, including CA180-031(NCT00337454); every 12 weeks (if on study >=6 months and <=2 years); every 24 weeks (if on study >2 years); at discontinuation
Population: All treated participants. Number of deaths represents all reported deaths, including after the study end. For AEs leading to discontinuation: 4 in CML-CP=1 insufficient effect (IE) +3 AEs in Participant Flow (PF); 7 in CML-AP/BP= 1 death + 5 AEs + 1 IE in PF; 4 in Ph+ALL=3 IE + 1AE in PF.
Measure: Number; unit: participants
Arm/Group | CML - Chronic Phase (CML-CP) | CML - Accelerated Phase and Blast Phase (CML-AP/BP) | Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL)
Number analyzed (Participants) | 30 | 11 | 13
participants
  AEs (symptoms/signs and laboratory abnormalities) | 30 | 11 | 13
  SAEs (symptoms/signs and laboratory abnormalities) | 13 | 9 | 11
  Deaths | 1 | 2 | 3
  AEs that led to discontinuation | 4 | 7 | 4

2. Secondary Outcome: Participants With Chronic Phase CML (CML-CP): Percentage of Participants With Cytogenetic Response
Description: Cytogenetic responses (CyR) are based on the percentage of Ph+ metaphases among at least 20 metaphase cells in each bone marrow (BM) sample. The criteria for cytogenetic responses are as follows. Best CyR is defined as the best response obtained at any time during the study. Major Cytogenetic Response (MCyR) = Complete Cytogenetic Response (CCyR; 0 Ph+ Cells in Metaphase in BM), plus Partial Cytogenetic Response (PCyR; 1 - 35 Philadelphia positive [Ph+] Cells in Metaphase in BM).
Time Frame: At baseline, every 24 weeks thereafter (including study CA180031/NCT00337454)
Population: Treated CML-CP participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- CML - Chronic Phase (CML-CP) Total: Imatinib resistant or intolerant CML-CP disease cohort who had completed the previous study (CA180031) phase I/II. The study drug was administered twice daily (BID). The starting dose level for this trial in each individual participant was the same dose level at the end of CA180031, allowed to modify within the range of 50 mg twice daily (BID) to 90 mg BID.
- CML - Chronic Phase (CML-CP) - Imatinib Resistant: Imatinib resistant CML-CP disease cohort who had completed the previous study (CA180031) phase II. The study drug was administered twice daily (BID). The starting dose level for this trial in each individual participant was the same dose level at the end of CA180031, allowed to modify within the range of 50 mg twice daily (BID) to 90 mg BID.
- CML - Chronic Phase (CML-CP) - Imatinib Intolerant: Imatinib intolerant CML-CP disease cohort who had completed the previous study (CA180031) phase II. The study drug was administered twice daily (BID). The starting dose level for this trial in each individual participant was the same dose level at the end of CA180031, allowed to modify within the range of 50 mg twice daily (BID) to 90 mg BID.
Arm/Group | CML - Chronic Phase (CML-CP) Total | CML - Chronic Phase (CML-CP) - Imatinib Resistant | CML - Chronic Phase (CML-CP) - Imatinib Intolerant
Number analyzed (Participants) | 30 | 11 | 12
Percentage of Participants
  Major cytogenetic response (MCyR) | 77 [57.7 to 90.1] | 61 [35.7 to 82.7] | 100 [73.5 to 100.0]
  Complete cytogenetic response (CCyR) | 63 [43.9 to 80.1] | 44 [21.5 to 69.2] | 92 [61.5 to 99.8]

3. Secondary Outcome: Participants With CML-Accelerated or Blast Phase (AP/BP): Percentage of Participants With Cytogenetic Response
Description: Cytogenetic responses (CyR) are based on the percentage of Ph+ metaphases among at least 20 metaphase cells in each bone marrow (BM) sample. The criteria for cytogenetic responses are as follows. Best CyR is defined as the best response obtained at any time during the study. Major Cytogenetic Response (MCyR) = Complete Cytogenetic Response (CCyR; 0 Ph+ Cells in Metaphase in BM), plus Partial Cytogenetic Response (PCyR; 1 - 35 Ph+ Cells in Metaphase in BM).
Time Frame: At baseline, every 12 weeks up to 2 years on study (including study CA180031/NCT00337454), every 24 weeks thereafter
Population: Treated CML-AP/BP participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- CML-AP/BP - Total Cohort: Imatinib resistant or intolerant CML-AP/BP disease cohort who had completed the previous study (CA180031) phase I/II. The study drug was administered twice daily (BID). The starting dose level for this trial in each individual participant was the same dose level at the end of CA180031, allowed to modify within the range of 50 mg twice daily (BID) to 90 mg BID.
- CML-AP/BP - Imatinib Resistant: Imatinib resistant CML-AP/BP disease cohort who had completed the previous study (CA180031) phase II. The study drug was administered twice daily (BID). The starting dose level for this trial in each individual participant was the same dose level at the end of CA180031, allowed to modify within the range of 50 mg twice daily (BID) to 90 mg BID.
- CML-AP/BP - Imatinib Intolerant: Imatinib intolerant CML-AP/BP disease cohort who had completed the previous study (CA180031) phase II. The study drug was administered twice daily (BID). The starting dose level for this trial in each individual participant was the same dose level at the end of CA180031, allowed to modify within the range of 50 mg twice daily (BID) to 90 mg BID.
Arm/Group | CML-AP/BP - Total Cohort | CML-AP/BP - Imatinib Resistant | CML-AP/BP - Imatinib Intolerant
Number analyzed (Participants) | 11 | 8 | 3
Percentage of Participants
  Major cytogenetic response (MCyR) | 27 [6.0 to 61.0] | 38 [8.5 to 75.5] | 0 [0 to 0]
  Complete cytogenetic response (CCyR) | 18 [2.3 to 51.8] | 25 [3.2 to 65.1] | 0 [0 to 0]

4. Secondary Outcome: Participants With Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL): Percentage of Participants With Cytogenetic Response
Description: as for outcome 3
Time Frame: At baseline, every 12 weeks up to 2 years on study (including study CA180031/NCT00337454), every 24 weeks thereafter
Population: Treated Ph+ ALL participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL) - Total Cohort: Ph+ ALL subjects with resistance or intolerance to past therapy and who had completed the previous study (CA180031) phase II. The study drug was administered twice daily (BID). The starting dose level for this trial in each individual participant was the same dose level at the end of CA180031, allowed to modify within the range of 50 mg twice daily (BID) to 90 mg BID.
- Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL) - Resistant: Ph+ ALL subjects with resistance to past therapy and who had completed the previous study (CA180031) phase II. The study drug was administered twice daily (BID). The starting dose level for this trial in each individual participant was the same dose level at the end of CA180031, allowed to modify within the range of 50 mg twice daily (BID) to 90 mg BID.
- Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL) - Intolerant: Ph+ ALL subjects with intolerance to past therapy and who had completed the previous study (CA180031) phase II. The study drug was administered twice daily (BID). The starting dose level for this trial in each individual participant was the same dose level at the end of CA180031, allowed to modify within the range of 50 mg twice daily (BID) to 90 mg BID.
Arm/Group | Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL) - Total Cohort | Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL) - Resistant | Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL) - Intolerant
Number analyzed (Participants) | 13 | 9 | 4
Percentage of Participants
  Major cytogenetic response (MCyR) | 54 [25.1 to 80.8] | 33 [7.5 to 70.1] | 100 [39.8 to 100.0]
  Complete cytogenetic response (CCyR) | 46 [19.2 to 74.9] | 22 [2.8 to 60.0] | 100 [39.8 to 100.0]

5. Secondary Outcome: Participants With CML-CP: Time to Complete Cytogenetic Response (CCyR)
Description: Cytogenetic responses (CyR) are based on the percentage of Ph+ metaphases among at least 20 metaphase cells in each bone marrow (BM) sample. Complete Cytogenetic Response (CCyR) = 0 Ph+ Cells in Metaphase in BM. Time to complete CCyR is defined as the time from first dose of dasatinib until measurement criteria are first met for CCyR, and is computed only for subjects whose best response is CCyR.
Time Frame: At baseline, every 24 weeks thereafter (including study CA180031/NCT00337454),
Population: Participants achieving CCyR
Measure: Median (Full Range); unit: Days
Arm/Group | CML - Chronic Phase (CML-CP)
Number analyzed (Participants) | 19
Days | 169 [83 to 841]

6. Secondary Outcome: Participants With CML-AP/BP and Ph+ ALL: Time to Complete Cytogenetic Response (CCyR)
Description: as for outcome 5
Time Frame: At baseline, every 12 weeks up to 2 years on study (including study CA180031/NCT00337454), every 24 weeks thereafter
Population: Participants achieving CCyR
Measure: Median (Full Range); unit: Days
Groups:
- Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL): Ph+ ALL subjects with resistance or intolerance to past therapy and who had completed the previous study (CA180031) phase II. The study drug was administered twice daily (BID). The starting dose level for this trial in each individual participant was the same dose level at the end of CA180031 (ie, 50mg, 70mg or 90mg BID on a continuous daily dosing schedule), allowed to modify within the range of 50 mg twice daily (BID) to 90 mg BID.
Arm/Group | CML - Accelerated Phase and Blast Phase (CML-AP/BP) | Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL)
Number analyzed (Participants) | 2 | 6
Days | 215 [93 to 337] | 82 [9 to 89]

7. Secondary Outcome: Participants With CML-CP: Duration of Complete Cytogenetic Response (CCyR)
Description: Cytogenetic responses (CyR) are based on the percentage of Ph+ metaphases among at least 20 metaphase cells in each bone marrow (BM) sample. Complete Cytogenetic Response (CCyR) = 0 Ph+ Cells in Metaphase in BM. Duration of CCyR was measured from the time measurement criteria are first met for CCyR until the first date of progressed disease (PD) or death. Subjects who neither relapsed nor died will be censored on the date of their last assessment.
Time Frame: At baseline, every 24 weeks thereafter (including study CA180031/NCT00337454)
Population: Participants achieving CCyR. Median duration of CCyR was not yet reached in the CML-CP group.
Measure: Median (Full Range); unit: Days
Arm/Group | CML - Chronic Phase (CML-CP)
Number analyzed (Participants) | 0

8. Secondary Outcome: Participants With CML-AP/BP and Ph+ALL: Duration of Complete Cytogenetic Response (CCyR)
Description: Cytogenetic responses (CyR) are based on the percentage of Ph+ metaphases among at least 20 metaphase cells in each bone marrow (BM) sample. Complete Cytogenetic Response (CCyR) = 0 Ph+ Cells in Metaphase in BM. Duration of CCyR was measured from the time measurement criteria are first met for CCyR until the first date of PD or death. Subjects who neither relapsed nor died will be censored on the date of their last assessment.
Time Frame: At baseline, every 12 weeks up to 2 years on study (including study CA180031/NCT00337454), every 24 weeks thereafter
Population: Participants achieving CCyR. Median duration of CCyR was not yet reached in the CML-AP/BP group.
Measure: Median (Full Range); unit: Days
Arm/Group | CML - Accelerated Phase and Blast Phase (CML-AP/BP) | Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL)
Number analyzed (Participants) | 0 | 6
Days |  | 96.5 [35 to 705]

9. Secondary Outcome: Participants With CML-CP: Time to Major Cytogenetic Response (MCyR)
Description: Major Cytogenetic Response (MCyR) = Complete Cytogenetic Response (CCyR; 0 Ph+ Cells in Metaphase in BM), plus Partial Cytogenetic Response (PCyR; 1 - 35 Ph+ Cells in Metaphase in BM). Time to MCyR was defined as the time from first dose of dasatinib until measurement criteria were first met for CCyR or PCyR (whichever status is recorded first).
Time Frame: At baseline, every 24 weeks thereafter (including study CA180031/NCT00337454)
Population: Time to MCyR was computed only for participants whose best response was CCyR or PCyR.
Measure: Median (Full Range); unit: Days
Arm/Group | CML - Chronic Phase (CML-CP)
Number analyzed (Participants) | 23
Days | 169 [83 to 1006]

10. Secondary Outcome: Participants With CML-AP/BP and Ph+ALL: Time to Major Cytogenetic Response (MCyR)
Description: as for outcome 9
Time Frame: At baseline, every 12 weeks up to 2 years on study (including study CA180031/NCT00337454), every 24 weeks thereafter
Population: Time to MCyR was computed only for participants whose best response was CCyR or PCyR.
Measure: Median (Full Range); unit: Days
Arm/Group | CML - Accelerated Phase and Blast Phase (CML-AP/BP) | Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL)
Number analyzed (Participants) | 3 | 7
Days | 85 [84 to 93] | 85 [5 to 96]

11. Secondary Outcome: Participants With CML-CP: Duration of Major Cytogenetic Response (MCyR)
Description: Major Cytogenetic Response (MCyR) = Complete Cytogenetic Response (CCyR; 0 Ph+ Cells in Metaphase in BM), plus Partial Cytogenetic Response (PCyR; 1 - 35 Ph+ Cells in Metaphase in BM). Duration of MCyR was measured from the time measurement criteria are first met for CCyR or PCyR (whichever status is recorded first) until the first date of progressive disease (PD) or death. Subjects who neither relapsed nor died were censored on the date of their last assessment.
Time Frame: At baseline, every 24 weeks thereafter (including study CA180031/NCT00337454)
Population: Duration of MCyR was computed for subjects whose best response was either CCyR or PCyR. Median duration of MCyR was not yet reached in the CML-CP arm.
Measure: Median (Full Range); unit: Days
Arm/Group | CML - Chronic Phase (CML-CP)
Number analyzed (Participants) | 0

12. Secondary Outcome: Participants With CML-AP/BP and Ph+ ALL: Duration of Major Cytogenetic Response (MCyR)
Description: as for outcome 11
Time Frame: At baseline, every 12 weeks up to 2 years on study (including study CA180031/NCT00337454), every 24 weeks thereafter
Population: Duration of MCyR was computed for subjects whose best response was either CCyR or PCyR. Median duration of MCyR was not yet reached in the CML-AP/BP arm.
Measure: Median (Full Range); unit: Days
Arm/Group | CML - Accelerated Phase and Blast Phase (CML-AP/BP) | Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL)
Number analyzed (Participants) | 0 | 7
Days |  | 85 [35 to 705]

13. Secondary Outcome: Participants With CML-CP: Percentage of Participants With Complete Hematologic Response (CHR)
Description: CHR=all of the following criteria: white blood cell count (WBC) ≤institutional upper limit of normal(ULN); platelets <450,000/mm³; no blasts or promyelocytes in peripheral blood; <5% myelocytes plus metamyelocytes in peripheral blood; peripheral blood basophils <20%; no extramedullary involvement.
Time Frame: baseline; every 4 weeks < 6 months on study (including study CA180031/NCT00337454), every 12 weeks >=6 months and <=2 years; every 24 weeks >2 years; at discontinuation
Population: Treated CML-CP participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | CML - Chronic Phase (CML-CP) Total | CML - Chronic Phase (CML-CP) - Imatinib Resistant | CML - Chronic Phase (CML-CP) - Imatinib Intolerant
Number analyzed (Participants) | 30 | 18 | 12
Percentage of Participants | 93 [77.9 to 99.2] | 89 [65.3 to 98.6] | 100 [73.5 to 100.0]

14. Secondary Outcome: Participants With CML-AP/BP: Percentage of Participants With Hematologic Response
Description: Major Hematologic Response=Complete Hematologic Response (CHR) or No Evidence of Leukemia (NEL). CHR=WBC <ULN; absolute neutrophil count (ANC) >1,000/mm3; platelets >100,000/mm3; no blasts or promyelocytes in peripheral blood; BM blasts ≤5%; <5% myelocytes + metamyelocytes in peripheral blood; <20% basophils in peripheral blood; no extramedullary involvement. NEL=(see Outcome Measure 15, below). Overall hematologic response (OHR)=best response of CHR, NEL or return to chronic phase (RTC).
Time Frame: baseline; every 4 weeks < 6 months on study (including study CA180031/NCT00337454); every 12 weeks >=6 months and <=2 years; every 24 weeks >2 years; at discontinuation
Population: Treated CML-AP/BP participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | CML-AP/BP - Total Cohort | CML-AP/BP - Imatinib Resistant | CML-AP/BP - Imatinib Intolerant
Number analyzed (Participants) | 11 | 8 | 3
Percentage of Participants
  Overall hematologic response (OHR) | 73 [39.0 to 94.0] | 75 [34.9 to 96.8] | 67 [9.4 to 99.2]
  Major hematologic response (MaHR) | 73 [39.0 to 94.0] | 75 [34.9 to 96.8] | 67 [9.4 to 99.2]
  Complete hematologic response (CHR) | 55 [23.4 to 83.3] | 75 [34.9 to 96.8] | 0 [0 to 0]

15. Secondary Outcome: Participants With Ph+ ALL: Percentage of Participants With Hematologic Response
Description: Major Hematologic Response=Complete Hematologic Response (CHR) or No Evidence of Leukemia (NEL). CHR=(see Outcome Measure 14, above). NEL=WBC ≤ULN; BM blasts ≤5%; no blasts or promyelocytes in peripheral blood; <5% myelocytes plus metamyelocytes in peripheral blood; <20% peripheral blood basophils; no extramedullary involvement; and at least 1 of the following: ANC ≥500/mm3 and <2000/mm3 or platelets ≥20,000/mm3 and <100,000/mm3. Overall hematologic response (OHR)=best response of CHR, NEL or return to chronic phase (RTC).
Time Frame: as for outcome 14
Population: Treated Ph+ ALL participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL) - Total Cohort | Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL) - Resistant | Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL) - Intolerant
Number analyzed (Participants) | 13 | 9 | 4
Percentage of Participants
  Overall hematologic response (OHR) | 69 [38.6 to 90.9] | 56 [21.2 to 86.3] | 100 [39.8 to 100.0]
  Major hematologic response (MaHR) | 46 [19.2 to 74.9] | 33 [7.5 to 70.1] | 75.5 [19.4 to 99.4]
  Complete hematologic response (CHR) | 15 [1.9 to 45.4] | 0 [0 to 0] | 50 [6.8 to 93.2]

16. Secondary Outcome: Time to Complete Hematologic Response (CHR) in Chronic Phase CML, Accelerated or Blast Phase CML, and Ph+ALL
Description: CHR=all of the following criteria: WBC ≤institutional upper limit of normal(ULN); platelets <450,000/mm³; no blasts or promyelocytes in peripheral blood; <5% myelocytes plus metamyelocytes in peripheral blood; peripheral blood basophils <20%; no extramedullary involvement. Time to CHR=time from first dose of dasatinib until the first day criteria for CHR are met provided they are confirmed 28 days later and was computed only for chronic phase CML subjects whose best response is CHR. Subjects who neither progressed nor died were censored at date of last hematologic assessment.
Time Frame: as for outcome 14
Population: Participants achieving CHR
Measure: Median (Full Range); unit: Days
Arm/Group | CML - Chronic Phase (CML-CP) | CML - Accelerated Phase and Blast Phase (CML-AP/BP) | Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL)
Number analyzed (Participants) | 29 | 6 | 2
Days | 12.5 [3 to 343] | 89 [57 to 307] | 98.5 [57 to 140]

17. Secondary Outcome: Duration of Complete Hematologic Response (CHR) in Chronic Phase CML, Accelerated or Blast Phase CML, and Ph+ALL
Description: Duration of CHR was computed only for chronic phase CML subjects whose best response is CHR. It was measured from the first day complete hematologic response criteria are met provided they are confirmed 28 days later until the date treatment is discontinued due to PD or death. Subjects who neither progressed nor died were censored on the date of their last hematologic assessment.
Time Frame: as for outcome 14
Population: Participants achieving CHR. Duration of CHR in the CML AP/BP arm has not yet been reached.
Measure: Median (Full Range); unit: Days
Arm/Group | CML - Chronic Phase (CML-CP) | CML - Accelerated Phase and Blast Phase (CML-AP/BP) | Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL)
Number analyzed (Participants) | 29 | 0 | 2
Days | 1160 [153 to 1310] |  | 373 [102 to 644]

18. Secondary Outcome: Time to Major Hematologic Response (MaHR) in Accelerated or Blast Phase CML, and Ph+ALL
Description: Major Hematologic Response=Complete Hematologic Response (CHR) or No Evidence of Leukemia (NEL; see Outcome Measures 14 and 15 for full definitions). Time to major hematologic response (MaHR)=time from first dose of dasatinib until the first day the measurement criteria for MaHR and is computed only for advanced diseases subjects whose best response is a major hematologic response. Subjects who neither progressed nor died were censored on the date of their last hematologic assessment.
Time Frame: as for outcome 14
Population: Participants achieving MaHR
Measure: Median (Full Range); unit: Days
Arm/Group | CML - Accelerated Phase and Blast Phase (CML-AP/BP) | Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL)
Number analyzed (Participants) | 8 | 6
Days | 45.5 [8 to 102] | 59 [9 to 151]

19. Secondary Outcome: Duration of Major Hematologic Response (MaHR) in Accelerated or Blast Phase CML, and Ph+ALL
Description: Major Hematologic Response (MaHR)=Complete Hematologic Response (CHR) or No Evidence of Leukemia (NEL; see Outcome Measures 14 and 15 for full definitions). Subjects who neither progressed nor died were censored on the date of their last hematologic assessment.
Time Frame: as for outcome 14
Population: Duration of MaHR was computed only for advanced diseases subjects whose best response is a MaHR and was measured from the first day MaHR criteria are met, provided they were confirmed 28 days later until the date of PD or death. Median Duration of MaHR was not yet reached in the CML-AP/BP arm.
Measure: Median (Full Range); unit: Days
Arm/Group | CML - Accelerated Phase and Blast Phase (CML-AP/BP) | Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL)
Number analyzed (Participants) | 0 | 6
Days |  | 102.5 [35 to 774]

20. Secondary Outcome: Time to Overall Hematologic Response (OHR) in Accelerated or Blast Phase CML, and Ph+ALL
Description: The overall hematologic response (OHR) rate is defined as the proportion of all treated subjects with a best response of major or minor hematologic response. Time to OHR = time from first dose of dasatinib until the first day measurement criteria are first met for hematologic response provided they were confirmed 28 days later. Subjects who neither progressed nor died were censored on the date of last hematologic assessment.
Time Frame: as for outcome 14
Population: OHR was computed only for subjects whose best response is CHR or MaHR or Minor HR (MiHR).
Measure: Median (Full Range); unit: Days
Arm/Group | CML - Accelerated Phase and Blast Phase (CML-AP/BP) | Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL)
Number analyzed (Participants) | 8 | 9
Days | 38.5 [8 to 68] | 13 [2 to 68]

21. Secondary Outcome: Duration of Overall Hematologic Response (OHR) in Accelerated or Blast Phase CML, and Ph+ALL
Description: The overall hematologic response (OHR) rate is defined as the proportion of all treated subjects with a best response of major or minor hematologic response. Subjects who neither progressed nor died were censored on the date of last hematologic assessment.
Time Frame: as for outcome 14
Population: Duration of OHR was computed only for participants whose best response was CHR or a MaHR or MiHR & was measured from the first day hematologic response criteria were met, provided they were confirmed 28 days later until the date of PD or death. Median duration of OHR in the CML-AP/BP arm was not yet reached.
Measure: Median (Full Range); unit: Days
Arm/Group | CML - Accelerated Phase and Blast Phase (CML-AP/BP) | Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL)
Number analyzed (Participants) | 0 | 9
Days |  | 104 [30 to 774]

22. Secondary Outcome: Participants With Detectable Mutations of RNA (mRNA) of BCR-ABL at Baseline and at Best Achievement
Description: Detectable BCR-ABL transcripts (b3a2, b2a2 or minor) >=2.0 log copy/micrograms RNA, as measured by real-time quantitative PCR (RQ-PCR) at baseline and best achievement post-dose.
Time Frame: At baseline, every 12 weeks up to 2 years on study (including study CA180031/NCT00337454), every 24 weeks thereafter, and at discontinuation
Population: Treated participants
Measure: Number; unit: participants
Arm/Group | CML - Chronic Phase (CML-CP) | CML - Accelerated Phase and Blast Phase (CML-AP/BP) | Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL)
Number analyzed (Participants) | 30 | 11 | 13
participants
  Baseline | 28 | 11 | 10
  Best Achievement | 12 | 7 | 6

23. Secondary Outcome: Status of Point Mutations of BCR-ABL at Baseline (BL) and End of Study (EOS)
Description: Point mutations of BCR-ABL detected or undetected in the Quantitative real-time PCR polymerase chain reaction (RQ-PCR) products
Time Frame: At baseline and discontinuation--the study period was extended until the launch of dasatinib in Japan, January 2009.
Population: Treated participants
Measure: Number; unit: participants
Arm/Group | CML - Chronic Phase (CML-CP) | CML - Accelerated Phase and Blast Phase (CML-AP/BP) | Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL)
Number analyzed (Participants) | 30 | 11 | 13
participants
  Undetectable at BL → Detectable at EOS | 1 | 1 | 7
  Detectable at BL → Detectable at EOS | 2 | 1 | 3
  Detectable at BL → Undetectable at EOS | 2 | 0 | 0
  Detectable at BL → Not Analyzed at EOS | 1 | 1 | 1

24. Secondary Outcome: Collection of Blood Samples for Pharmacokinetic Analysis of Dasatinib Twice Daily (BID) That Will Contribute to Population Pharmacokinetic Modeling
Description: Blood samples for pharmacokinetic analysis of Dasatinib BID that will contribute to population pharmacokinetic modeling were collected.
Time Frame: At any visit of later than Day 7, draw sample(s) at pretreatment trough (within 1 hour prior to dosing) or between 3 hours following treatment and prior to the next dose
Population: There was no individual PK analysis done for this study; analyses were integrated and evaluated as a part of population PK of this drug.
Measure: Number; unit: participants
Arm/Group | CML - Chronic Phase (CML-CP) | CML - Accelerated Phase and Blast Phase (CML-AP/BP) | Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- All Treated Participants: Imatinib resistant or intolerant CML-CP disease cohort, Imatinib resistant or intolerant CML-AP/BP disease cohort, and Ph+ ALL subjects with resistance or intolerance to past therapy. The study drug was administered twice daily (BID). The starting dose level for this trial in each individual participant was the same dose level at the end of CA180031 (ie, 50mg, 70mg or 90mg BID on a continuous daily dosing schedule), allowed to modify within the range of 50 mg twice daily (BID) to 90 mg BID.
Arm/Group | All Treated Participants
Serious Adverse Events (participants affected / at risk) | 33/54
Other Adverse Events (participants affected / at risk) | 54/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Treated Participants (N=54)
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial tachycardia (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Anal fistula (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Periodontitis (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 3
Malaise (General disorders) | 1
Therapeutic response decreased (General disorders) | 1
Disease progression (General disorders) | 1
Pneumonia (Infections and infestations) | 6
Enteritis infectious (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Perianal abscess (Infections and infestations) | 1
Pseudomembranous colitis (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 2
Brain herniation (Injury, poisoning and procedural complications) | 1
Drug toxicity (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Haemothorax (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Platelet count decreased (Investigations) | 4
Haemoglobin decreased (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Haematocrit decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Red blood cell count decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Tumour lysis syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Blast cell crisis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haemorrhage (Nervous system disorders) | 3
Convulsion (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Brain mass (Nervous system disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Haematoma (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Treated Participants (N=54)
Anaemia (Blood and lymphatic system disorders) | 23
Febrile neutropenia (Blood and lymphatic system disorders) | 6
Neutropenia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Cardiomegaly (Cardiac disorders) | 5
Palpitations (Cardiac disorders) | 5
Pericardial effusion (Cardiac disorders) | 4
Sinus bradycardia (Cardiac disorders) | 3
Hypothyroidism (Endocrine disorders) | 3
Eyelid oedema (Eye disorders) | 10
Conjunctival haemorrhage (Eye disorders) | 8
Conjunctival hyperaemia (Eye disorders) | 5
Vision blurred (Eye disorders) | 4
Conjunctivitis (Eye disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 32
Nausea (Gastrointestinal disorders) | 21
Constipation (Gastrointestinal disorders) | 18
Vomiting (Gastrointestinal disorders) | 16
Stomatitis (Gastrointestinal disorders) | 15
Abdominal pain (Gastrointestinal disorders) | 7
Toothache (Gastrointestinal disorders) | 7
Abdominal distension (Gastrointestinal disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 6
Cheilitis (Gastrointestinal disorders) | 5
Gingivitis (Gastrointestinal disorders) | 5
Haematochezia (Gastrointestinal disorders) | 5
Abdominal pain lower (Gastrointestinal disorders) | 4
Gingival bleeding (Gastrointestinal disorders) | 4
Haemorrhoids (Gastrointestinal disorders) | 4
Stomach discomfort (Gastrointestinal disorders) | 4
Dental caries (Gastrointestinal disorders) | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3
Gingival swelling (Gastrointestinal disorders) | 3
Pyrexia (General disorders) | 27
Malaise (General disorders) | 23
Oedema (General disorders) | 18
Oedema peripheral (General disorders) | 9
Face oedema (General disorders) | 7
Pain (General disorders) | 7
Chest pain (General disorders) | 5
Chills (General disorders) | 5
Chest discomfort (General disorders) | 3
Fatigue (General disorders) | 3
Hypothermia (General disorders) | 3
Seasonal allergy (Immune system disorders) | 3
Nasopharyngitis (Infections and infestations) | 29
Folliculitis (Infections and infestations) | 8
Pharyngitis (Infections and infestations) | 6
Bronchitis (Infections and infestations) | 5
Gastroenteritis (Infections and infestations) | 4
Infection (Infections and infestations) | 4
Influenza (Infections and infestations) | 3
Excoriation (Injury, poisoning and procedural complications) | 7
Transfusion reaction (Injury, poisoning and procedural complications) | 3
Wound (Injury, poisoning and procedural complications) | 3
Neutrophil count decreased (Investigations) | 46
Platelet count decreased (Investigations) | 42
White blood cell count decreased (Investigations) | 41
Blood lactate dehydrogenase increased (Investigations) | 39
Lymphocyte count decreased (Investigations) | 39
Aspartate aminotransferase increased (Investigations) | 35
Alanine aminotransferase increased (Investigations) | 34
Blood creatine phosphokinase increased (Investigations) | 30
Gamma-glutamyltransferase increased (Investigations) | 25
Haematocrit decreased (Investigations) | 25
Haemoglobin decreased (Investigations) | 25
Red blood cell count decreased (Investigations) | 24
Blood phosphorus decreased (Investigations) | 24
Blood albumin decreased (Investigations) | 23
Protein urine present (Investigations) | 23
White blood cell count increased (Investigations) | 22
Protein total decreased (Investigations) | 20
Blood alkaline phosphatase increased (Investigations) | 19
Weight increased (Investigations) | 18
Blood urine present (Investigations) | 17
Weight decreased (Investigations) | 17
Blood uric acid increased (Investigations) | 16
CD4 lymphocytes decreased (Investigations) | 16
Blood creatinine increased (Investigations) | 12
Blood urea increased (Investigations) | 10
Urinary sediment abnormal (Investigations) | 10
Reticulocyte count decreased (Investigations) | 9
Urobilin urine present (Investigations) | 9
Blood potassium decreased (Investigations) | 8
Electrocardiogram QT corrected interval prolonged (Investigations) | 8
Glucose urine present (Investigations) | 8
Protein urine (Investigations) | 8
Blood bilirubin increased (Investigations) | 7
Blood magnesium increased (Investigations) | 7
Blood potassium increased (Investigations) | 7
C-reactive protein increased (Investigations) | 7
Liver function test abnormal (Investigations) | 7
Lymphocyte count increased (Investigations) | 6
Neutrophil count increased (Investigations) | 5
CD4 lymphocytes increased (Investigations) | 5
Blood pressure increased (Investigations) | 4
Blood sodium decreased (Investigations) | 4
Prothrombin time prolonged (Investigations) | 4
Reticulocyte count increased (Investigations) | 4
Platelet count increased (Investigations) | 4
Activated partial thromboplastin time prolonged (Investigations) | 3
Blood chloride decreased (Investigations) | 3
Eosinophil count increased (Investigations) | 3
Urine ketone body present (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 12
Decreased appetite (Metabolism and nutrition disorders) | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 14
Back pain (Musculoskeletal and connective tissue disorders) | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 4
Joint swelling (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Headache (Nervous system disorders) | 26
Dizziness (Nervous system disorders) | 7
Hypoaesthesia (Nervous system disorders) | 6
Dysgeusia (Nervous system disorders) | 5
Insomnia (Psychiatric disorders) | 7
Haematuria (Renal and urinary disorders) | 3
Gynaecomastia (Reproductive system and breast disorders) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 27
Erythema (Skin and subcutaneous tissue disorders) | 8
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 8
Purpura (Skin and subcutaneous tissue disorders) | 8
Acne (Skin and subcutaneous tissue disorders) | 7
Petechiae (Skin and subcutaneous tissue disorders) | 5
Eczema (Skin and subcutaneous tissue disorders) | 4
Skin exfoliation (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 3
Rash papular (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 5
Hypotension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.